CLINICAL TRIAL: NCT06205888
Title: To Compare the Clinical Application of 18F-LNC1007 (18F-FAPI-RGD) and 18F-FDG PET/CT in Tumor Diagnosis, Staging and Recurrence Detection
Brief Title: To Compare the Clinical Application of 18F-LNC1007 Injection PET/CT and 18F-FDG PET/CT
Acronym: 18F-LNC1007
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Jinling Hospital, China (Other)
Responsible Party: Principal Investigator, Jiang Wu, archiater, Jinling Hospital, China
Other Study IDs: 18F-LNC1007
Record Dates: First submitted 2024-01-04; First posted 2024-01-16 (Actual); Last update posted 2024-01-16 (Actual); Status verified 2024-01

CONDITIONS: Tumour
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Compare 18F-LNC1007 injection (18F-FAPI-RGD) PET/CT and 18F-FDG PET/CT imaging: This is a prospective, controlled, open-label (with blind members), single-center clinical trial to evaluate the diagnostic efficacy and safety of 18F-LNC1007 injection PET/CT for suspected tumor or tumor initial staging, recurrence monitoring, etc.
  Interventions: Other: 18F-LNC1007（18F-FAPI-RGD） PET/CT和18F-FDG PET/CT

INTERVENTIONS:
Other: 18F-LNC1007（18F-FAPI-RGD） PET/CT和18F-FDG PET/CT — Eligible subjects will receive 18F-LNC1007 (18F-FAPI-RGD) PET/CT and 18F-FDG PET/CT examinations within 1 week (the interval between the two examinations shall not exceed 7 days, and the scanning parameters, scanning range, image reconstruction methods, etc., shall be consistent). That is, with 18F-LNC1007 (18F-FAPI-RGD) PET/CT time as D0, 18F-FDG PET/CT examination can accept data from D1 to D7

SUMMARY:
To evaluate the safety of 18F-LNC1007 injection in the diagnosis of suspected tumor, initial stage, or recurrence monitoring; to explore the biological distribution of 18F-LNC1007 injection in patients; To compare the diagnostic efficacy of 18F-LNC1007 injection PET/CT versus 18F-FDG PET/CT imaging in patients with tumor with clinical suspicion, initial stage, or recurrence monitoring.

DETAILED DESCRIPTION:
This is a prospective, controlled, open-label (with blind members), single-center clinical trial to evaluate the diagnostic efficacy and safety of 18F-LNC1007 injection PET/CT for suspected tumor or tumor initial staging, recurrence monitoring, etc.

ELIGIBILITY:
Inclusion Criteria:

* (1) Age ≥18 years old; (2) Clinically suspected or confirmed tumor patients; (3) As judged by doctors, the expected survival time is 3 months; (4) Voluntarily sign informed consent; (5) Willing and able to follow the research protocol; (6) The subject must be able to lie on the scanning bed for at least 1 hour.

Exclusion Criteria:

* (1) known allergic history to 18F-LNC1007 injection; (2) Patients who cannot tolerate intravenous drug administration (such as needle fainting and blood fainting history); (3) Those who are not suitable for PET/CT and other imaging examinations or cannot complete them due to special reasons, including claustrophobia and radiophobia; (4) pregnant and lactating women; (5) Workers who are exposed to radiation for a long period of time; (6) serious diseases of the heart, kidney, lung, blood vessel, nervous system, mental system, immune deficiency diseases and hepatitis/cirrhosis; (7) Participating in other interventional clinical trials within 1 month before screening; (8) Patients undergoing chemotherapy, immunotherapy or molecular targeted therapy; (9) There are other circumstances that the researcher considers inappropriate to participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A patient with a clinically suspected or confirmed tumor
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
To evaluate the sensitivity and specificity of 18F-LNC1007 (18F-FAPI-RGD) PET/CT at the patient level compared with 18F-FDG PET/CT; | 3 months
  To evaluate the sensitivity and specificity of 18F-LNC1007 (18F-FAPI-RGD) PET/CT at the patient level compared with 18F-FDG PET/CT;

SECONDARY OUTCOMES:
Compare the difference of the uptake of imaging agent between 18F-LNC1007 (18F-FAPI-RGD) and 18F-FDG injection in tumor lesions or metastases | 3 months
  Compare the difference of the uptake of imaging agent between 18F-LNC1007 (18F-FAPI-RGD) and 18F-FDG injection in tumor lesions or metastases

OTHER OUTCOMES:
The type, incidence, and severity of adverse events were graded using the National Cancer Institute Standard for Common Terminology for Adverse Events (NCI CTCAE) V5.0 standard | 3 months
  The type, incidence, and severity of adverse events were graded using the National Cancer Institute Standard for Common Terminology for Adverse Events (NCI CTCAE) V5.0 standard